CLINICAL TRIAL: NCT06623019
Title: Study of the Validity and Reliability of Two Digital Dynamometers in Older People
Acronym: SOVARDDIOP
Status: Completed | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Associate Professor, University of Salamanca
Other Study IDs: USalamancaValidityDinamometers
Record Dates: First submitted 2024-09-19; First posted 2024-10-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sarcopenia; Old Age; Debility; Frailty
Keywords: Muscle Strength Dynamometer; Hand Strength; aged; Muscle Fatigue; Jamar
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Device 1, Device 2 and Jamar®: As this is a validation study, both criterion, inter-observer and intra-observer validation will be performed. Initially, three repetitions will be performed with each device, leaving between 3 and 5 minutes of rest between devices. 20-30 minutes later, the same process will be repeated but with another researcher giving the orders (interobserver reliability). A few days later the same process is repeated with the first investigator (intra-observer reliability). No person will receive any treatment.
  Interventions: Diagnostic Test: Validation and reliability

INTERVENTIONS:
Diagnostic Test: Validation and reliability — As this is a cross-sectional validation study, there is no intervention.

SUMMARY:
It is a cross-sectional, randomized, and single-center study with a duration of 6 months. The study will follow the STROBE guidelines for cross-sectional studies and CONSORT 2024. The main objective is to evaluate the validity and reliability of two devices in measuring grip strength and muscle fatigability in community-dwelling older adults.The study will include community-dwelling older adults of both sexes over 60 years of age.

DETAILED DESCRIPTION:
Design: It is a cross-sectional, randomized, and single-center study with a duration of 6 months. The study will follow the STROBE guidelines for cross-sectional studies and CONSORT 2024. The main objective is to evaluate the validity and reliability of the Device 1 and Device 2 devices in measuring grip strength and muscle fatigability in community-dwelling older adults.

It will be carried out in two stages: In a first moment the criterion and interobserver validity will be assessed and in a second moment the intraobserver validity. Participants will be randomly assigned to one of the 6 arms to follow different orders of the devices (Device 1, Device 2 or Jamar).

Population: community-dwelling older adults of both sexes over 60 years of age.

Procedures: The investigators will schedule each participant for the initial assessment day. Using a table of random numbers, they will be assigned one of the arms. All participants have previously read, signed and given their written informed consent. An interview will be conducted in which age, sex and medication will be collected; an anthropometric and functional assessment will be performed. The functional tests include the 30-second squat test and grip strength tests using the Jamar, Device 1 and Device 2. Three repetitions will be performed with each device, allowing 30 seconds between repetitions and 3 to 5 minutes between devices. After 20 minutes the test will be repeated again on the devices for interobserver validation. 5 to 10 days later, tester 1 will repeat the grip test with the same effort to assess intraobserver reliability.

Sample size: Similar studies validating grip strength devices compared to the Jamar showed an excellent correlation (ICC > 0.90). With an estimated ICC of 0.90 ± 0.05 and an alpha risk of 5%, 348 participants are required for the training study.

Variables: Sociodemographic (age, sex, hand dominance, number of medication types), anthropometric (height, weight, BMI and SMI), strength and fatigability (total number of repetitions in 30sCS, maximal grip strength (HGS), fatigue resistance (FR) and grip work (GW)) and device preference.

Statistical analysis: Maximal strength and fatigability will be analyzed by means of means, standard deviations and statistical tests. Concordance between devices will be assessed using the Kappa coefficient and the Bland-Altman concordance index. ROC curves will be used to determine sensitivity and specificity, and data will be analyzed by gender. Results will be considered statistically significant if p < 0.05, and IBM SPSS Statistics v28.0 will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults of both sexes over 60 years of age.

Exclusion Criteria:

* Those who do not understand the orders given to them by the researcher or present an obvious advanced state of dementia.
* Those people who have amputation in one of the two upper limbs or who cannot perform manual grasping for any reason.
* Those who have had an episode of pain in one of the hands during the week prior to the measurement.
* Those who, due to any illness, prevent or contraindicate maximum resistance exercises.
* Any other cause that the research team assesses that may affect the results.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling older adults of both sexes over 60 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
2. Hand grip test | 2 weeks
  Measurement of hand grip strength using a hand-held dynamometer. Values shall be recorded with all three devices.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | 2 weeks
  Is a mathematical ratio that associates the mass and the size of an individual BMI = weight / height ^2
4. Appendicular Skeletal Muscle mass Index (SMI) | 2 weeks
  Is a mathematical ratio that associates the muscle mass and the size of an individual SMI = appendicular muscle mass / height ^2
30 seconds chair stand test (30sCS) | 2 weeks
  Test that measures the number of times you perform the maximum number of squats on a chair in 30 seconds. The more squats the better functionally.
Fatigue resistance (FR) | 2 weeks
  Time taken to lose 50% of the maximum recorded grip strength.
Grip work (GW) | 2 weeks
  Value resulting from multiplying the maximum grip force by the fatigue strength by 0,75. It is measured in watts.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Polo-Ferrero, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain